CLINICAL TRIAL: NCT03420573
Title: Clinical Profile of Parkinson's Disease in Patients With Hepatitis C Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Shaimaa El-Jaafary, Lecturer of Neurology, Kasr El Aini Hospital
Other Study IDs: KAMDUPDHC
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is association between Hepatitis C and Parkinson's Disease as shown from previous studies. The clinical profile and natural history is not fully studied yet. We aim at studying the clinical characteristics of Parkinson's Disease in patients with hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with history of Parkinson's Disease and Hepatitis C infection.

Exclusion Criteria:

* Advanced liver cirrhosis.
* Patients with hepatic failure.
* Symptoms of Parkinson's plus syndrome.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease patients with hepatitis C infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Score of UPDRS | 2 years
  Severity of Motor and non motor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa I. El-Jaafary, MD, Study Director — Director of Kasr Alainy Movement Disorders Unit KAMDU

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous Demographic data ,severity of symptoms, score results

REFERENCES:
- [Background] Pakpoor J, Noyce A, Goldacre R, Selkihova M, Mullin S, Schrag A, Lees A, Goldacre M. Viral hepatitis and Parkinson disease: A national record-linkage study. Neurology. 2017 Apr 25;88(17):1630-1633. doi: 10.1212/WNL.0000000000003848. Epub 2017 Mar 29. PMID 28356465
- [Background] Kim JM, Jang ES, Ok K, Oh ES, Kim KJ, Jeon B, Jo HJ, Ki M, Jeong SH. Association between hepatitis C virus infection and Parkinson's disease. Mov Disord. 2016 Oct;31(10):1584-1585. doi: 10.1002/mds.26755. No abstract available. PMID 27549922
- [Background] Golabi P, Otgonsuren M, Sayiner M, Arsalla A, Gogoll T, Younossi ZM. The Prevalence of Parkinson Disease Among Patients With Hepatitis C Infection. Ann Hepatol. 2017 May-Jun;16(3):342-348. doi: 10.5604/16652681.1235476. PMID 28425403